CLINICAL TRIAL: NCT03048604
Title: A Multicentre, Prospective, Open-label, Non-randomized, Single Arm Treatment Study to Assess the Safety, Performance and Initial Efficacy Trends of the Genio(TM) Bilateral Hypoglossal Nerve Stimulation System for the Treatment of Obstructive Sleep Apnoea.
Brief Title: BiLAteral Hypoglossal Nerve Stimulation for Treatment of Obstructive Sleep Apnoea (BLAST OSA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nyxoah S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BLAST OSA
Record Dates: First submitted 2017-02-07; First posted 2017-02-09 (Estimated); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Obstructive Sleep Apnea of Adult

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Genio(TM) system therapy (Experimental)
  Interventions: Device: Genio(TM) bilateral hypoglossal nerve stimulation system

INTERVENTIONS:
Device: Genio(TM) bilateral hypoglossal nerve stimulation system — Subjects will be consented, enrolled and eligibility criteria checked. If the subject is eligible, subject will proceed with the Genio(TM) implant implantation. Four (4) weeks after implantation, the implant will be activated and the subject will be assessed at 1 month plus 1 week, 2, 3, 4 and 6 month(s) after implantation.

SUMMARY:
The study is designed as a prospective, open-label, multicentre, non-randomized, single arm treatment study to assess the safety, performance and initial efficacy trends of the GenioTM System in patients with Obstructive Sleep Apnoea (OSA).

ELIGIBILITY:
Main Inclusion Criteria:

* Body mass index ≤32 kg/m2
* Patients who do not tolerate or do not accept positive airway pressure (PAP) treatments.
* Obstructive apnoea-hypopnea index (AHI) of 20-60 events/hour

Main Exclusion Criteria:

* Unable or incapable of providing informed written consent
* Unwilling or incapable of returning to all follow-up visits and sleep studies, including evaluation procedures and filling out questionnaires
* Significant co-morbidities making the patient unable or inappropriate to participate in the trial

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2018-09-10 (Actual); Study Completion 2018-09-10 (Actual)

PRIMARY OUTCOMES:
Safety (Incidence of serious device-related adverse events) | 6-months post implantation
  Incidence of serious device-related adverse events
Performance | 6-months post implantation
  Change from baseline to 6-month post implantation in the apnoea-hypopnea index (AHI)

CONTACTS AND LOCATIONS:
Overall Officials: Valérie Attali, Dr., Principal Investigator — La Pitié Salpêtrière, Paris
Locations (3):
- Hollywood Private UWA Centre for Sleep Science Facility, Nedlands, Perth, Australia
- La Pitié Salpêtrière - Paris, Paris, France
- Royal National Throat, Nose and Ear Hospital - London, London, United Kingdom

REFERENCES:
- [Derived] Eastwood PR, Barnes M, MacKay SG, Wheatley JR, Hillman DR, Nguyen XL, Lewis R, Campbell MC, Petelle B, Walsh JH, Jones AC, Palme CE, Bizon A, Meslier N, Bertolus C, Maddison KJ, Laccourreye L, Raux G, Denoncin K, Attali V, Gagnadoux F, Launois SH. Bilateral hypoglossal nerve stimulation for treatment of adult obstructive sleep apnoea. Eur Respir J. 2020 Jan 9;55(1):1901320. doi: 10.1183/13993003.01320-2019. Print 2020 Jan. PMID 31601716